CLINICAL TRIAL: NCT00164268
Title: Ke Ala Lokahi Demonstration Project for the Early Intervention and Prevention of Sexual and Domestic Violence Among Racial and Ethnic Populations
Brief Title: Ke Ala Lokahi Demonstration Project for Sexual and Domestic Violence Prevention
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCIPC-11249; US4/CCU919035-02
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2007-09-10 (Estimated); Status verified 2007-09

CONDITIONS: Domestic Violence
Keywords: Intimate partner violence; Sexual violence; Cultural intervention; Native Hawaiian

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Ke Ala Lokahi (Native Hawaiian cultural intervention)

SUMMARY:
The purpose of the project is to examine the efficacy of a culturally-based intervention, compared to standard agency services, in enhancing self-care among Native Hawaiian women and decreasing IPV/SV perpetration and related factors among Native Hawaiian men.

DETAILED DESCRIPTION:
Turning Point for Families in Hilo, Hawaii is developing, implementing, and evaluating a culturally-based intervention using Native Hawaiian values, beliefs, and practices to address intimate partner and sexual violence among Native Hawaiian perpetrators and victims/survivors.

ELIGIBILITY:
Inclusion Criteria:

* Men and women self-identified as Native Hawaiian referred for agency services due to intimate partner or sexual violence

Exclusion Criteria:

* See above. No other exclusion criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 2002-10; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Subsequent incidents of intimate partner or sexual violence for up to 2 years post-intervention

SECONDARY OUTCOMES:
Attitudes, behaviors, and cultural identity assessed at 3-months, 6-months, and 15-months following treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Linda Slutter, Principal Investigator — Turning Point for Families
Locations (1):
- Turning Point for Families, Hilo, Hawaii, United States